CLINICAL TRIAL: NCT06752447
Title: A Phase I Clinical Study of Safety, Tolerability, Pharmacokinetic/pharmacodynamic Characteristics and Initial Efficacy of LNF2007 Monotherapy in Patients with Advanced Solid Tumors
Brief Title: A Phase I Study OfLNF2007 Monotherapy in Patients with Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTP-LNF2007-001
Record Dates: First submitted 2024-12-22; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Advanced Solid Tumors (Phase 1)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LNF2007 monotherapy (Experimental)
  Interventions: Drug: LNF2007

INTERVENTIONS:
Drug: LNF2007 — LNF2007，9 dose groups:0.2μg/kg、1μg/kg、5μg/kg、20μg/kg、60μg/kg、120μg/kg、240μg/kg、360μg/kg、540μg/kg（0.2~5μg/kg for "accelerated titration", and i3+3 ramp-up starting from 20μg/kg dose group），IV, infusion time 60min±10min, Q4W, until disease progression 、intolerable toxicity or other reasons to stop treatment, the longest administration to 2 years, whichever occurs first.

SUMMARY:
A non-randomized, open-ended, phase I dose-escalation and dose-expansion study was designed to evaluate the safety, tolerability, antitumor efficacy, PK and immunogenic characteristics of LNF2007 in patients with advanced solid tumors

DETAILED DESCRIPTION:
A non-randomized, open-ended, phase I dose-escalation and dose-expansion study was designed to evaluate the safety, tolerability, antitumor efficacy, PK and immunogenic characteristics of LNF2007 in patients with advanced solid tumors. This study is divided into dose escalation stage and dose extension stage.

A total of 9 dose groups were designed in the dose escalation phase. The dose expansion phase is planned to be conducted in two dose groups (determined by discussion between the investigator and sponsor based on available trial data), enrolling approximately 20 participants at each dose. According to the results of dose escalation phase, the pre-excitation dose of dose extension phase is designed.

ELIGIBILITY:
Inclusion Criteria:

* Study participants must meet all of the following inclusion criteria to be enrolled in the study:

  1. Age ≥18 years old, gender unlimited;
  2. United States Eastern Oncology Consortium (ECOG) physical strength score 0-1;
  3. Expected survival ≥12 weeks;
  4. Patients with advanced solid tumors confirmed histologically or cytologically (gastric cancer, pancreatic cancer, and cholangiocarcinoma are preferred) who have failed after adequate standard treatment, or who lack standard treatment options (standard treatment is defined as the standard treatment guidelines that have been agreed in the country (if applicable) or the standard treatment status in the country); Standard treatment failure is defined as disease progression or tumor recurrence or metastasis during or after treatment, or intolerance);
  5. Agree to provide archived tumor tissue specimens or fresh tissue specimens within 2 years of the primary or metastatic lesion (to explore the characteristics of biomarkers in tumor tissue); If the subject is unable to provide a tumor tissue sample, the participant can be enrolled after evaluation by the investigator, provided that other inclusion criteria are met.
  6. There is at least one evaluable tumor lesion according to RECIST V1.1;
  7. Tumor tissue samples were confirmed to be Claudin18.2 positive by immunohistochemical (IHC) detection, and positive was defined as ≥1+ by IHC detection (only applicable to patients in the dose escalation phase of 60μg/kg or above and in the dose expansion phase);
  8. Adequate organ function before the first administration of the test drug (no blood components, cell growth factors, whitening drugs, platelet enhancing drugs, etc., have been used within 14 days before the first administration) 1.Absolute neutrophil count ≥1.5×109/L; 2.Platelet ≥100×109/L; 3.Hemoglobin ≥90g/L; 4.Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN (for liver cancer or liver metastasis, ≤5×ULN); Total bilirubin (TBIL) ≤1.5×ULN (liver cancer or liver metastasis, ≤3×ULN); 5. Serum creatinine (Cr) ≤1.5×ULN, creatinine clearance (CLcr) ≥50mL/min when Cr > 1.5×ULN (CLcr was calculated using Cockcroft-Gault equation); 6.Activated partial thromboplastin time (APTT) ≤1.5×ULN, International Normalized ratio (INR) ≤1.5×ULN.
  9. Understand and voluntarily sign informed consent.

Exclusion Criteria:

* Study participants with any of the following were not eligible for the study:

  1. Received any antitumor therapy within 4 weeks prior to the first use of the investigational drug or within 5 half-lives of the drug (whichever is shorter);
  2. Had undergone major organ surgery (excluding needle biopsy) or significant trauma within 4 weeks prior to the first use of the trial drug, or required elective surgery during the trial;
  3. Received systemic corticosteroid (systemic corticosteroid equivalent to prednisone >10mg daily) or other immunosuppressive therapy within 2 weeks prior to the first use of the experimental drug;
  4. Prior to first administration of the investigational drug, all reversible adverse effects of previous antitumor therapy did not return to CTCAE v5.0 rating ≤1, excluding alopecia (any grade) and ≤2 peripheral sensory neuropathy or other toxicities deemed by the investigators to be of no safety risk;
  5. Received dual antibody or CAR-T drug therapy targeting Claudin18.2 within 3 months before the first use of the experimental drug;
  6. have an active autoimmune disease and have had systemic systemic treatment within 3 months prior to the first use of the trial drug;
  7. Patients with clinical symptoms of central nervous system metastasis and other evidence of uncontrolled central nervous system metastasis were judged by the investigators to be unsuitable for inclusion; Any meningeal metastases;
  8. Subjects with a known history of severe hypersensitivity to other monoclonal antibodies or intravenous gamma globulin, and a known history of hypersensitivity or hypersensitivity to LNF2007 components;
  9. have a severe systemic active infection that currently requires systemic anti-infection therapy;
  10. Patients with active gastrointestinal bleeding or other gastrointestinal diseases deemed unsuitable for inclusion by researchers as having high risk factors for gastrointestinal bleeding, such as active gastrointestinal perforation requiring clinical intervention, pyloric obstruction, complete or incomplete intestinal obstruction, etc.;
  11. There are clinical symptoms of pleural effusion, pericardial effusion or ascites requiring frequent drainage (≥1 time/month);
  12. Impaired heart function or suffering from major cardiovascular and cerebrovascular diseases, including but not limited to:

  <!-- -->

  1. myocardial infarction, unstable angina pectoris, cerebrovascular accident, acute or persistent myocardial ischemia, symptomatic heart failure (grade 2 or higher according to the New York Heart Association Functional Scale), symptomatic or poorly controlled arrhythmia, or any arterial thromboembolism event in the six months prior to initial administration;
  2. History of deep vein thrombosis, pulmonary embolism, or other serious thromboembolism within 3 months prior to the first dose;
  3. aortic aneurysm, aortic dissection aneurysm, internal carotid artery stenosis and other major vascular diseases that may be life-threatening or require surgery within 6 months;
  4. Previous history of myocarditis and cardiomyopathy;
  5. Left ventricular ejection fraction (LVEF) < 50%; 13) Patients currently suffering from interstitial lung disease or pulmonary fibrosis, pneumoconiosis, radiation pneumonia, severe impairment of lung function, etc., which may interfere with the detection and management of suspected drug-related pulmonary toxicity; 14) Hepatitis B patients (if HBsAg and/or HBcAb positive and HBV-DNA≥200IU/ml (or 1000cps/ml)); Hepatitis C patients (HCV antibody positive and HCV-RNA testing indicates viral replication); Syphilis screening positive (specific antibody test positive, non-specific antibody test negative and combined with clinical judgment confirmed as inactive infection), known HIV positive history or HIV screening positive; 15) The patient is known to have a history of psychotropic substance abuse, alcohol abuse or drug use; 16) Pregnant or lactating women, female subjects of childbearing age, or male subjects with partners of women of childbearing age who did not consent to contraception during the study period and within 6 months after the last study drug treatment; 17) Two or more malignancies in the 5 years prior to the first dose. With the exception of early stage malignancies that have been cured (carcinoma in situ or stage I tumours), such as carcinoma in situ of the cervix, basal cell or squamous cell skin cancer that has been adequately treated; 18)Patients who were not suitable for enrollment according to the judgment of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of LNF2007 treatment-emergent adverse events | Through up to approximately 30 days following last dose of LNF2007
  Incidence and severity of AEs and specific laboratory abnormalities graded according to NCI-CTCAE, v5.0
Occurrence of dose-limiting toxicity (DLT) | Within 28 days after first target dose
  DLTs will include Grade 4 neutropenia, anemia, thrombocytopenia, ≥ Grade 3 Febrile neutropenia ，Grade 5 toxicity and other Grade 3 non-hematological toxicity etc
The maximum tolerated dose and/or the recommended phase II dose of LNF2007 | the first 3 weeks of treatment
  Dose Finding

IPD SHARING:
Plan to Share IPD: No